CLINICAL TRIAL: NCT01499186
Title: The Effect of 6 Months of Local Vibration Training of the Thigh and Hip on Muscle Strength, Muscle Mass, Bone Density, Bone Structure and Functionality in Institutionalized Elderly.
Brief Title: The Effect of 6 Months of Local Vibration Training in Institutionalized Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ML7837
Record Dates: First submitted 2011-12-19; First posted 2011-12-26 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2013-12

CONDITIONS: Osteoporosis; Sarcopenia
Keywords: Local vibration, elderly, bone, muscle, functionality
MeSH Terms: conditions — Osteoporosis; Sarcopenia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): There will be no participation in a training program. The control group will perform all measurements.
- Intervention group (Experimental): The subjects of the vibration group will be subjected to local vibration training by the use of custom-made cylindrical vibrators. These subjects will perform all measurements.
  Interventions: Other: Local Vibration

INTERVENTIONS:
Other: Local Vibration — The subjects of the vibration group will be subjected to local vibration training by the use of custom-made cylindrical vibrators which will be placed on the hip and thigh. The subjects will apply the vibrations by themselves and they will learn how to follow the pre-programmed training program. Training sessions take place 5 times a week, during one year. The physiotherapist and the research assistant will attend the training session 1x/week. Training parameters will vary during the year to create a variable stimulus (frequency 40-80Hz and G-force 0.5-5g). The intervention group will perform all measurements.
  Other Names: Local vibration of muscle and bone
  Arms: Intervention group

SUMMARY:
This randomized controlled intervention study in institutionalized elderly investigates the effect of 6 months of local vibration therapy applied on the thigh and hip on muscle strength, muscle mass, bone density, and functionality.

DETAILED DESCRIPTION:
As the world population ages, osteoporosis (skeletal fragility) and sarcopenia (decline in muscle mass and muscle strength) are becoming increasingly important public health concerns. Both osteoporosis and sarcopenia contribute to an increased fall risk and an increased number of hip and vertebral fractures. Clearly, the clinical and economic consequences of osteoporosis and sarcopenia, and the resulting falls and fractures, call for major efforts to search for efficient and feasible interventions to prevent or reverse bone and muscle loss. The present project is intended to partly meet this need.

Whole Body Vibration (WBV) training might be an efficient training method. During WBV the subject stands on a platform that generates vertical sinusoidal vibrations. These mechanical stimuli are transmitted to the body where they stimulate the bone and reflexive muscle contractions will be generated. In previous studies performed by the same group, the investigators found that WBV training (frequency 30-40Hz, peak acceleration 3-10g) can be seen as an efficient alternative for strength training, both in the young sedentary as well as in the elderly population. Additionally, the investigators were able to show that 6 months vibration training in elderly females resulted in a net benefit of about 1.5% in bone mineral density of the hip compared with controls. Finally, the investigators have recently shown that long-term vibration training results in an increase of quadriceps muscle mass.

From the above it appears that vibration therapy could be a plausible candidate as an efficient combination therapy for elderly subjects at risk for osteoporosis and sarcopenia and, by implication, the therapy might help to reduce the number of falls and fractures. However, many questions regarding vibration as a therapy still need to be answered in order to optimize both the efficacy and safety of its application. The application methods of vibration therapy should be optimized to be applicable in a broader range of subjects as well as to deliver the stimuli more targeted to specific regions of interest. Whole body vibration in its present form (subjects standing on a vibrating platform) is inadequate for a large part of the elderly population (e.g., subjects with osteoarthritis at the knee, wheelchair bound subjects, bedridden subjects). Additionally, the transmission of the vibration stimulus from the feet to the hip during WBV is probably insufficient to provoke optimal adaptations at this level. Delivering the vibration stimuli locally (i.e. more targeted) at those regions at risk for fractures or in need for muscle strengthening might be an efficient alternative application method.

The main aim of this pilot research is to obtain data that should allow the investigators to optimize the efficacy and safety of the vibration excitation pattern as well as to optimize the application method. With the ageing of the world population and the predicted rise in fall and fracture rates, appropriate strategies to combat muscle and bone loss will have far reaching implications in containing future health care expenditure for the elderly and in reducing the need for institutionalized care.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Above 65 years of age;
* Institutionalized in a nursing home, service flat or cloistered community;
* Not on bone-active agents;
* Approval for participation in the study after a medical screening by a doctor. The general practitioner will also be contacted for approving the participation of the patient;
* Signed informed consent.

Exclusion Criteria:

* Musculoskeletal disease;
* Terminal illness, recent myocardial infarction or unstable cardiovascular conditions;
* Participation in resistance training during the past 24 months;
* Metallic implants (e.g. prothesis);

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Bone mineral density hip (change in bone mineral density hip) | baseline and after 6 months
  Bone mineral density of the total hip will be determined by dual - energy x - ray absorptiometry (Hologic, Waltham, MA, USA).

SECONDARY OUTCOMES:
Functionality (change in functionality) | baseline and 6 months
  Functionality will be determined by the modified Physical Performance Test (mPPT). Additionally, the number of falls during the study period and their circumstances will be identified using Fall calendars.
Physical performance (change in physical performance) | baseline and 6 months
  Physical performance will be assessed by the "shuttle walk test" which is a standardized incremental field walking test that provokes a symptom limited maximal performance
Muscle mass (change in muscle mass) | baseline and 6 months
  Muscle mass of the upper leg will be determined by a multislice CT-scan (Siemens Sensation 16) which delivers axial slices of the right upper leg. The midpoint between the medial edge of the greater trochanter and the intercondyloid fossa of the patella was determined, and subsequently a 2 mm-thick axial image (1 mm above and 1 mm below this midpoint) was further analyzed. This procedure was repeated 3 cm above and 3 cm below the midpoint. Muscle tissue area was segmented by using standard Hounsfield Units ranges for skeletal muscle (0-100).
Muscle strength and muscle power (change in muscle strength and power) | baseline and 6 months
  Muscle strength and muscle power of the knee extensors will be measured on an isokinetic dynamometer. Static and dynamic muscle strength will be recorded unilaterally on the Biodex Medical System 3 dynamometer. A standard protocol will be performed twice: isometric strength (120 °, 90° en 30°), isotonic strength with 40%, 20% and 1% of the isometric maximum and isokinetic strength by 60°/s, 180°/s en 240°/s.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Verschueren, PhD, Prof, Principal Investigator — KU Leuven
Locations (1):
- Faculty of Kinesiology and Rehabilitation Sciences, Leuven, Vlaams Brabant, Belgium

REFERENCES:
- [Derived] Tankisheva E, Bogaerts A, Boonen S, Delecluse C, Jansen P, Verschueren SM. Effects of a Six-Month Local Vibration Training on Bone Density, Muscle Strength, Muscle Mass, and Physical Performance in Postmenopausal Women. J Strength Cond Res. 2015 Sep;29(9):2613-22. doi: 10.1519/JSC.0000000000000895. PMID 25992656